CLINICAL TRIAL: NCT01417871
Title: ABC Program in Patients With Metabolic Syndrome
Status: Completed | Type: Observational
Sponsor: University of Magdeburg (Other)
Responsible Party: Claus Luley, University Magdeburg
Other Study IDs: abcmetsyn1
Record Dates: First submitted 2011-08-15; First posted 2011-08-16 (Estimated); Last update posted 2011-08-16 (Estimated); Status verified 2010-02

CONDITIONS: Weight Reduction in Patients With Metabolic Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples for parameter of lipid metabolism
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- case goup: Lifestyle counseling, ABC program
- control group: usual care

SUMMARY:
Aims: We evaluate the efficacy of the "Active Body Control (ABC) Program" for weight reduction in patients with metabolic syndrome.

Methods: The ABC program combines telemonitoring of the physical activity with a low-calorie diet also preferring carbohydrates with low glycemic indexes. In this 12-month, randomized, clinical trial 60 patients will be treated according to the ABC program and 60 control patients will receive standard therapy.

ELIGIBILITY:
Inclusion Criteria:

* metabolic syndrome

Exclusion Criteria:

* tumor cachexia

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with metabolic syndrome
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2010-02; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
weight reduction | 12 month

SECONDARY OUTCOMES:
incidence of metabolic syndrome | 12 month

CONTACTS AND LOCATIONS:
Locations (1):
- University Magdeburg, Magdeburg, Germany